CLINICAL TRIAL: NCT04838392
Title: Effectiveness and Safety of the RIGHTEST Continuous Glucose Monitoring System for Blood Glucose Management in Persons With Diabetes Mellitus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bionime Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: US-312-01
Record Dates: First submitted 2021-03-29; First posted 2021-04-09 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Diabetes Mellitus; Type 1 Diabetes; Type 2 Diabetes
Keywords: Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Masking Description: All information as provided by CGM system will be masked from subjects and study team during the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- CGM System (Experimental): Blood draw and glucose challenge will be performed to evaluate the performance of the CGM system compared to reference measurements during the in in-clinic visits.
  Interventions: Device: RIGHTEST Continuous Glucose Monitoring System

INTERVENTIONS:
Device: RIGHTEST Continuous Glucose Monitoring System — RIGHTEST Continuous Glucose Monitoring System

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of the RIGHTEST Continuous Monitoring (CGM) System in adult population with diabetes mellitus.

DETAILED DESCRIPTION:
This is a prospective, open-label, randomized, multicenter, single-arm pivotal study without control groups in up to 150 adult subjects with type 1 or type 2 diabetes mellitus who will be enrolled at 12 investigational sites in the United States.

All subjects are required to wear 1 Sensor on the back of each upper arm for up to 15 days (up to 360 hours) and participate in 4 in-clinic visits. All subjects will have frequent venous blood draws to evaluate the blood glucose reference measurements in each in-clinic visit and collect accurate information against a laboratory reference method.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years and older
* Subjects must have a diagnosis of type 1 or type 2 diabetes mellitus
* Subjects must be available to participate in all clinical sessions with the following parameters:
* Subject must be willing to wear 1 sensor on each upper arm simultaneously.
* Subjects must be willing to have their glucose levels manipulated in each in-clinic visit.
* Subjects must be able to follow the instructions provided to him/her by the study site and perform all study tasks as specified by the protocol.
* Subjects must be willing and able to provide signed written consent.
* Subjects must be able to speak, read and write English.

Exclusion Criteria:

* Known allergy and not able to tolerate to medical grade tape adhesive.
* Presence and unresolved of extensive skin changes/diseases at sensor wear site(s) that preclude wearing the sensor(s) on skin
* Subjects who have or are female of child-bearing potential age:

  * Has a positive pregnancy screening test
  * That plans to become pregnant during the course of study.
* Diagnosed with hemophilia or any other bleeding disorders
* Acute or chronic kidney disease
* Currently managed by dialysis or anticipating initiating dialysis during the course of study.
* Current or know history of coronary artery or cardiovascular disease that is not stable with medical management thromboembolic disease.
* Any condition that, in the opinion of the Investigator, would interfere with their participation in the study or pose excessive risk to study staff.
* Prior to enrollment, subject has had:

  * Severe hypoglycemia within past 6 months.
  * History of Diabetic Ketoacidosis (DKA) within the past 6 months,
  * History of a seizure disorder within the last 6 month
  * Hypoglycemia unawareness.
  * Severe diabetes related complications.
  * Required or scheduled to have a Magnetic Resonance Imagining (MRI) scan, Computed Tomography (CT) scan, or diathermy during the study wear period.
  * Plans to donate blood during the course of the study
  * Insulin-dependent type 2 subjects that receive sodium-glucose cotransporter 2 inhibitor (SGLT2 inhibitor) treatment[14]
  * Hematocrit (Hct) level lower than the normal reference range
  * Weight less than 110 pounds (50 kg)
* Participated in another clinical trial within 2 weeks prior to screening
* Unable to follow clinical protocol for the duration of the study or is otherwise deemed unacceptable to participate in the study per the Investigator's clinical judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
RIGHTEST Continuous Glucose Monitoring System Performance | 15 days
  The CGM System performance will be primarily evaluated in terms of point and trend accuracy of RIGHTEST™ CGM System continuous interstitial glucose measurements compared to the reference method.

SECONDARY OUTCOMES:
To investigate the RIGHTEST Glucose Monitoring System other system performance and safety | 15 days
  The secondary objective is to investigate other system performance by comparing the CGM System readings to the reference method. System performance includes the point and the trend accuracy, the precision of the CGM system, the stability of the CGM system across the wear period, and the glucose event alert function. The safety of RIGHTEST CGM will be examined through the number and percentage of subjects experiencing adverse events and examined through symptoms related to the Sensor insertion site.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Lakeview Clinical Research, Guntersville, Alabama
  - Novak Clinical Research, Tucson, Arizona
  - Hope Clinical Research LLC, Canoga Park, California
  - AMCR Institute, Escondido, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Infinite Clinical Trials, Morrow, Georgia
  - L-MARC Research Center, Louisville, Kentucky
  - Research Integrity, LLC., Owensboro, Kentucky
  - Scott Research,Inc, Laurelton, New York
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Oregon Health, Portland, Oregon
  - The Research Center of the Upstate, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No